CLINICAL TRIAL: NCT03854994
Title: A Phase I Clinical Trial of Anti-CD19 Chimeric Antigen Receptor With Synthetic Biology Optimizing Nano-vector T Cells Injection for Subjects With Relapsed/Refractory/High-risk B-cell Lymphoma and B-cell Acute Lymphoblastic Leukemia
Brief Title: CD19 CAR-T Cell Therapy for Relapsed/Refractory B-cell Lymphoma and B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Collaborators: KAEDI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201707202
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: B Cell Lymphoma; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 CAR-T Cells Injection (Experimental): Dosage form：injection Dosage:1-5x10^6/kg, 70ml/time, The CAR-T cells will be administered by i.v. injection over 20-30 minutes Frequency: total one time
  Interventions: Biological: Anti-CD19 CAR-T Cells Injection

INTERVENTIONS:
Biological: Anti-CD19 CAR-T Cells Injection — Autologous genetically modified anti-CD19 CAR transduced T cells
  Other Names: KD-019 CAR-T cells Injection

SUMMARY:
The primary objective of this study is to evaluate the safety and clinical activity of anti-CD19 Chimeric Antigen Receptor T cells (KD-019 CAR-T)infusion in the treatment of relapsed/refractory B-cell Lymphoma and B-cell acute lymphoblastic leukemia （B-ALL）.

DETAILED DESCRIPTION:
The investigators designed an KD-019 Chimeric Antigen Receptor(CAR) with FMC63 single-chain antibody fragment (Scfv). This CAR has a CD8 hinge and transmembrane domains and a 4-1BB costimulatory domain; T cells expressing this CAR release relatively low levels of cytokines. Subjects with relapsed/refractory CD19-positive B-cell Lymphoma and B-ALL can participate if all eligibility criteria are met. Subjects receive chemotherapy prior to the infusion of KD-019 CAR-T cells. After the infusion, subjects will accept follow-up for side effects and effect of KD-019 CAR-T cells by the sponsor. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the Informed Consent Document;
2. 18 Years and older, Male and female;
3. Pathologically and histologically confirmed CD19 + B cell tumors; Patients currently have no effective treatment options, such as chemotherapy or relapse after hematopoietic stem cell transplantation; Or patients voluntarily choose transfusion of anti-CD19 CAR-T cells as the first treatment program;

B-cell tumors / lymphomas and B-cell acute lymphoblastic leukemia include the following four types:

1. B-cell acute lymphoblastic leukemia;
2. Indolent B-cell lymphomas;
3. Aggressive B-cell lymphoma; 4、 Subjects:

(1) Residual lesions remain after treatment; (2) Not suitable for Hematopoietic stem cell transplantation (auto/allo-HSCT); (3) Relapse after Complement receptor 1 (CR1) and unsuitable for HSCT; (4) Patients with high risk factors; (5) Relapse or no remission after hematopoietic stem cell transplantation or cell immunotherapy.

5、 Have measurable or evaluable tumor foci; 6、 Liver, kidney and cardiopulmonary functions meet the following requirements:

1. Serum glutamic pyruvic transaminase (ALT) and serum glutamic oxaloacetic transaminase (AST) <3 ×upper limit of normal (ULN);
2. Total bilirubin ≤34.2μmol/L;
3. Serum creatinine<220μmol/L;
4. Baseline oxygen saturation≥95%;
5. Left ventricular ejection fraction（LVEF）≥40%. 7、 Subjects who did not receive Chemotherapy, Radiotherapy, Immunotherapy (immunosuppressive drugs) or other treatment within 4 weeks prior to enrollment; Relevant toxicity≤1 grade before enrollment (except for low toxicity such as hair loss); 8、Peripheral superficial venous blood flow is smooth, which can meet the needs of intravenous drip; 9、Clinical performance status of eastern cancer cooperation group (ECOG) score ≤2，Expected survival≥3 months;

Exclusion Criteria:

1. Pregnant (urine/blood pregnancy test positive) or lactating women;
2. Planned pregnancy during treatment or within 1 year after treatment, or a male subject whose partner plans pregnancy within 1 year of their cell transfusion;
3. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 year after enrollment;
4. Active or uncontrollable infection within four weeks prior to enrollment;
5. Patients with active hepatitis B/C;
6. HIV-infected patients;
7. Severe autoimmune or immunodeficiency disorders;
8. Patients are allergic to macromolecule drugs such as antigens or cytokines;
9. Subjects participated in other clinical trials within 6 weeks before enrollment;
10. Systematic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Mental illness;
12. Drug abuse/addiction;
13. The investigators consider other conditions unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with severe cytokine release syndrome(CRS) as a Measure of Safety and Tolerability. | 0 to 14 days post infusion
  The severe CRS post KD-019 CAR-T cells treatment will be evaluated and the maximum tolerated dose will be determined.
Copies numbers of CAR in peripheral blood (PB) | 1 year post infusion
  Copies numbers of CAR in peripheral blood (PB)

SECONDARY OUTCOMES:
Overall survival | 2 years post infusion
  For all subjects, overall survival refers to the period from being included in the test group to death caused by any reason
Duration of Response after administration | 2 years post infusion
  Duration of Response after administration
Progress Free Survival after administration | 2 years post infusion
  Progress Free Survival after administration

CONTACTS AND LOCATIONS:
Overall Officials: Peixian Zhang, Study Director — Kunming Yan'an Hospital
Locations (1):
- Kunming Yan'an Hospital, Oncology Department, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided